CLINICAL TRIAL: NCT04050501
Title: Non-invasive Vagus Nerve Stimulation in Acute Ischemic Stroke
Acronym: NOVIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government); ElectroCore INC (Industry)
Responsible Party: Principal Investigator, Marieke JH Wermer, MD, Professor Doctor, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL64702.058.18
Record Dates: First submitted 2019-08-05; First posted 2019-08-08 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Ischemic Stroke
Keywords: Brain infarction; Brain ischemia; Vagus nerve stimulation; Penumbra
MeSH Terms: conditions — Ischemic Stroke; Brain Infarction; Brain Ischemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: PROBE design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- non-invasive Vagus Nerve Stimulation (Active Comparator): non-invasive Vagus Nerve Stimulation on top of best medical practice
  Interventions: Device: non-invasive Vagus Nerve Stimulator
- Standard Care (No Intervention): Best medical practice alone

INTERVENTIONS:
Device: non-invasive Vagus Nerve Stimulator — Two stimulations of two minutes each will be applied in the neck every 15 minutes in the first 3 hours. Thereafter two stimulations will be applied every 8 hours over the next 5 days or until discharge, whichever occurs first. The stimulation side in the neck will be the radiological side of the stroke.
  Arms: non-invasive Vagus Nerve Stimulation

SUMMARY:
The main objective of the study will be to investigate whether treatment with non-invasive vagus nerve stimulation (nVNS) on top of best medical practice in acute ischemic stroke patients results in less infarct growth in the penumbra and smaller infarct volumes compared with those of patients not treated with nVNS. The study will be a prospective randomized clinical trial with blinded outcome assessment (PROBE design). 150 patients will be randomized to nVNS with the gammaCore Sapphire™ device on top of best medical practice versus best medical practice alone (including intravenous thrombolysis and/or thrombectomy if indicated). If patients are randomized to nVNS, two stimulations of two minutes each will be applied in the neck every 15 minutes in the first 3 hours. Thereafter two stimulations will be applied every 8 hours over the next 5 days or until discharge, whichever occurs first. The stimulation side in the neck will be the radiological side of the stroke. The primary endpoint will be the final infarct volume on MRI scan on day 5 of patients treated with nVNS compared with those of patients not treated with VNS.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke
* NIHSS ≥1
* Perfusion deficit on the admission CTP scan; the penumbra must comprise at least 1/3 of the total ischemic area (ischemic core and penumbra)
* The infarct has to comprise the anterior circulation
* Treatment has to start <12 hours after stroke onset
* Patients or their representatives need to give their informed consent

Exclusion Criteria:

* A life expectancy of less than three months
* mRS >2 prior to admission
* Contra-indication for contrast CT
* Contra-indications for VNS:

  * An active implantable medical device such as a pacemaker, deep brain stimulator, or any implanted electronic device
  * Symptomatic stenosis or dissection of the carotid artery (in these patients the other side will be stimulated unless a significant stenosis on the other side is present as well)
  * Structural abnormality e.g. lymphadenopathy, previous surgery or abnormal anatomy (in these patients the other side will be stimulated)
  * Metal cervical spine hardware or metallic implant near the stimulation site
  * Cervical vagotomy (in these patients the other side will be stimulated)
  * Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Infarct volume | On day 5
  Final infarct volume on MRI scan

SECONDARY OUTCOMES:
Feasibility of nVNS | On day 5
  Reached if more than 75% of the nVNS treated patients complete treatment for five days or until discharge
Tolerability of nVNS | On day 5
  Reached if less than 10% of the patients treated with nVNS has to abort treatment due to side effects
NIHSS (National Institutes of Health Stroke Scale) on day 5 | On day 5
  The scale runs from 0-42 and quantifies stroke severity
Clinical outcome (modified Rankin Scale, mRS) on day 90 | On day 90
  The scale runs from 0-6 and quantifies disabilities:
  0 - No symptoms
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities
  3. - Moderate disability. Requires some help, but able to walk unassisted
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent
  6. - Dead
Occurrence of seizures in the first 90 days | On day of admission, day 5 and day 90
  This will be asked to patients and their physician
Occurrence of headache in the first 90 days | On day of admission, day 5 and day 90
  A questionnaire will be taken adjusted from van Os et al., neurology 2016
Occurrence of depression in the first 90 days | On day 90
  HADS (Hospital Anxiety and Depression Scale) questionnaire will be taken. The scale runs from 0-21 and defines the risk of having a depression
Quality of life after 90 days | On day 90
  EQ5D-5L questionnaire will be taken. This questionnaire defines a health index based on different questions
Cognitive status on day 90 | On day 90
  TICS questionnaire will be taken. This questionnaire can assess cognitive status.
Penumbra recovery | On day 3
  Proportion of patients in whom <50% of the penumbra turned into ischemic core on non-contrast CT
Blood-brain barrier measurement | On day 3
  Degree of blood-brain barrier leakage on day three measured with CTP

CONTACTS AND LOCATIONS:
Overall Officials: Marieke JH Wermer, MD PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Derived] van der Meij A, van Walderveen MAA, Kruyt ND, van Zwet EW, Liebler EJ, Ferrari MD, Wermer MJH. NOn-invasive Vagus nerve stimulation in acute Ischemic Stroke (NOVIS): a study protocol for a randomized clinical trial. Trials. 2020 Oct 26;21(1):878. doi: 10.1186/s13063-020-04794-1. PMID 33106174

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-05-06): https://cdn.clinicaltrials.gov/large-docs/01/NCT04050501/SAP_000.pdf